CLINICAL TRIAL: NCT05241314
Title: Intergenerational Trauma in War-affected Families: Promoting Adolescent Adjustment Through a Family Mindfulness-based Intervention
Brief Title: FMBI With War-affected Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00011195
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Family Mindfulness-based Intervention in War-affected Families; Intergenerational Trauma; War-Related Trauma
MeSH Terms: conditions — Historical Trauma; War-Related Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 2 Youth (Experimental): One randomly selected index youth per participating Karen family. Community health worker interventionists (CHWI) will deliver 7 weeks of home-based intervention with optional post-intervention focus groups to examine the feasibility of the community-based participatory research approach and intervention delivery by CHWIs.
  Interventions: Behavioral: Learning to BREATHE
- Phase 2 Caregivers/Adults (Experimental): Maternal and paternal caregivers (if present) of participating Karen family. Community health worker interventionists (CHWI) will deliver 7 weeks of home-based intervention with optional post-intervention focus groups to examine the feasibility of the community-based participatory research approach and intervention delivery by CHWIs.
  Interventions: Behavioral: After Deployment Adaptive Parenting Tools (ADAPT)

INTERVENTIONS:
Behavioral: Learning to BREATHE — A 6 session group-based intervention targeting adolescent mindfulness. The adapted and merged intervention will be delivered to individual families (home-based) in twice-weekly sessions over a 7-week period by two community health worker interventionists.
  Arms: Phase 2 Youth
Behavioral: After Deployment Adaptive Parenting Tools (ADAPT) — A 14 session group-based mindful parenting intervention originally developed to increase emotion regulation among military caregivers with young children and improve youth adjustment. The adapted and merged intervention will be delivered to individual families (home-based) in twice-weekly sessions over a 7-week period by two community health worker interventionists.
  Arms: Phase 2 Caregivers/Adults

SUMMARY:
This study has two central research questions: 1) Is implementing a family mindfulness-based intervention with war-affected immigrant families through community based participatory research methods feasible?; and 2) Does the intervention demonstrate preliminary improvements in the social and behavioral health of war-affected caregivers and youth by addressing patterns of behavior that potentiate intergenerational trauma? The objective in the proposed study is to use Community Based Participatory Research strategies to test the feasibility and acceptability of a mindfulness-based intervention for Karen refugee families living post-resettlement in the United States. A key focus in this phase of the pilot will be intervention adaptation and establishing fidelity monitoring and quality improvement procedures through which the PI and community health worker interventionists are trained and evaluated in the delivery of the intervention.

DETAILED DESCRIPTION:
Intergenerational trauma is a major public health problem impacting war-affected families. The investigators' specific research contribution will test the feasibility of a 7-week family mindfulness-based intervention addressing key mechanisms central to the health of war-affected families. The significance of this contribution is tied to the conceptual understanding that caregivers uniquely influence the ways in which their children process trauma, experience stressful events, and thrive socially, behaviorally and physically. The responses of youth, in turn, affect the well-being of their parents. Left unaddressed, intergenerational trauma will continue to negatively impact the health and life course of immigrant youth and families. Collectively, this contributes to: higher burden of unaddressed mental and physical health disturbances in caregivers and youth; disruptions in family systems and community structures that negatively impact educational achievement and other indicators of youth adjustment; and increased exposure to familial and community violence. If a mindfulness-based intervention delivered directly to war-affected families in their homes can demonstrate improvements in the behavioral and social health effects of war trauma experienced by caregivers and their youth, then this study has the potential to offer a novel, effective approach to disrupting the generational impacts of war on war-affected families. The study will engage mothers, fathers, and youth to address intergenerational trauma fully. The investigators will establish plans for collaborative dissemination with WellShare International in phase I of the Clinical Translational Research Service pilot award, including academic dissemination (presentation and publication) as well as dissemination of results among key stakeholders and community members.

ELIGIBILITY:
Inclusion Criteria:

* Adult inclusion criteria:

  * Above the age of 18
  * Karen refugees resettled to the United States greater than one year prior to enrollment
  * Caregiving responsibility for at least one child between the ages of 11 and 18
  * Reported primary or secondary torture or war trauma exposure, based on assessments conducted during UMN IRB STUDY00000729
  * Participation in UMN IRB STUDY00000729 and having agreed to be contacted for future research
* Youth inclusion criteria:

  * Ages 11 to 18
  * Living in the home with the primary caregivers
  * Considered a dependent of the primary caregivers (still in high school or transitioning from school to workforce, not married and/or raising their own children - will take individual youth circumstances into consideration individually to make a determination of dependence)

Exclusion Criteria:

* Self-reported or study team observed severe or unstable mental or physical illness such as acute psychosis, presence or risk of safety concerns, and/or a physical disability or illness, which prevents the potential participant from engaging in the study activities. Youth will be excluded if screening is positive for PTSD. Caregivers will not be excluded if mental health screening is positive for PTSD/severe depression.
* Nonbiological caregiving relationships with child
* If one member of the family declines to participate in the initial enrollment, the family will be excluded. If the randomly selected index youth declines to participate, we will open enrollment to other youth in the family that meet the inclusion criteria.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hoffman, PHD, MPH, MSN, RN, Principal Investigator — University of Minnesota School of Nursing
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1 described in the IRB protocol was for intervention adaptation only and not human subjects research. We did not record individual outcomes or baseline information but used the information to inform implementation in phase 2. This record is for phase 2 part of the study and not phase 1.
Groups:
- Caregiver: Engaged Karen refugee caregivers in 14 session mindful parenting intervention Intervention: ADAPT
- Youth: Engaged Karen adolescent youth in 6 session mindfulness intervention Intervention: Learning to BREATHE
Period: Overall Study
Arm/Group | Caregiver | Youth
Started | 14 | 11
Completed | 10 | 10
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregiver | Youth | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 11 | 11
  Between 18 and 65 years | 14 | 0 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 11 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Youth Adjustment
Description: Strengths and Difficulties Questionnaire (SDQ I/S). A 25-item youth behavioral screening questionnaire, Total difficulties score: generated by summing scores from all the scales except prosocial scale, Range 0-40. Higher score, higher adjustment challenges
Time Frame: 3 months
Population: This outcome measure only pertains to the youth group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 0 | 10
units on a scale |  | -2.3 [-8.1 to 3.5]

2. Primary Outcome: Mindfulness
Description: Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). A 12-item assessment of mindfulness as a single construct. Items 2, 6, and 7 reverse-scored. After reversals, sum values for items 1-12. Sum of all values reflect greater mindful qualities.
  The range of the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) is 12-48. It is a 12-item scale where each item is rated on a 1-4 Likert scale, with higher scores indicating greater mindfulness.
Time Frame: 3 months
Population: This outcome measure only pertains to the youth group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 0 | 10
units on a scale |  | 0.5 [-0.9 to 1.9]

3. Primary Outcome: Youth Trauma History, PTSD Screening
Description: UCLA Brief Screen for Child/Adolescent Trauma and PTSD (UCLA-B). A 11-item (+2 open ended) evaluation of trauma history and PTSD symptoms for identifying at-risk cases. A cutoff score of 35 is highly sensitive and specific for detecting a diagnosis of PTSD. Higher score, higher burden of PTSD symptoms
  UCLA brief trauma screen: This was a screening tool used to establish the eligibility of youth participants. This was not included in the analysis.
  Each item on the scale is rated on a 0-4 scale, with higher scores signifying greater symptom severity, range 0-44. The FACES instrument is not scored based on a range, as described.
Time Frame: 3 months
Population: This outcome measure only pertains to the youth group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 0 | 10
units on a scale |  | 0.6 [-1.67 to 2.87]

4. Primary Outcome: Emotion Regulation
Description: Emotion Regulation Skills Questionnaire (ERSQ). A 27-item assessment of emotion regulation skills described in the ART model. Calculated mean of all questions. Higher score indicates better Emotion Regulation.
  The Emotion Regulation Skills Questionnaire (ERSQ) is a 27 item scale that uses a 5-point Likert scale for each item, 0 (not at all) to 4 (almost always), with a total score range of 0-108.
Time Frame: 3 months
Population: This outcome measure only pertains to the youth group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 0 | 10
units on a scale |  | -1.1 [-3.47 to 1.27]

5. Primary Outcome: Parent Mental Health Distress
Description: Karen Mental Health Screener - Brief (KMHS-B). 5-item measure developed to screen for mental distress associated with MDD and PTSD. Possible score ranges for five items 0-15. For clinical use, clinical cut score of 4.
  Higher score, higher burden of PTSD symptoms. Used cut score to refer
Time Frame: 3 months
Population: Measure only pertains to the caregiver group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 9 | 0
units on a scale | 0.44 [-2.30 to 3.19] |

6. Secondary Outcome: Physical Health Status
Description: Cohen-Hoberman Inventory of Physical Symptoms (CHIPS). A 33-item assessment of perceived burden from physical symptoms. Total score generated by summing items. Range 0-132. Higher score, higher burden of physical symptoms
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 9 | 10
units on a scale | 0.047 [-0.139 to 0.23] | 0.013 [-0.057 to 0.083]

7. Secondary Outcome: Family Functioning
Description: Family Adaptability and Cohesion Scale IV (FACES). A 42-item assessment of cohesion and flexibility. Dividing the average of the balanced scales (Cohesion and Flexibility) by the average of the unbalanced scales (Rigid, Enmeshed, Chaotic and Rigid). The higher the ratio score the more balanced the family system.
  Each item on the scale is rated on a 0-4 scale, with higher scores signifying greater symptom severity, range 0-44. The FACES instrument is not scored based on a range, as described.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 9 | 10
units on a scale | 0.002 [-0.006 to 0.009] | 0.003 [-0.001 to 0.008]

8. Secondary Outcome: Emotion Regulation
Description: Emotion Regulation Skills Questionnaire (ERSQ). A 27-item assessment of emotion regulation skills described in the ART model.
  ESRQ - 27 items, each scored 0-4, range 0-108, higher scores mean higher emotion regulation. Total scores used, no subscales. Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) has a range of scores from 12 to 48, each of the 12 items is rated on a 4-point Likert scale (from "Rarely/Not at all" to "Almost Always") with higher scores indicating greater mindfulness.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 9 | 10
units on a scale | 0.062 [-0.436 to 0.559] | 0.137 [-0.428 to 0.702]

9. Secondary Outcome: Mindfulness
Description: Cognitive and Affective Mindfulness Scale- Revised (CAMS-R). A 12-item assessment of mindfulness as a single construct. Items 2, 6, and 7 reverse-scored. After reversals, sum values for items 1-12. Sum of all values reflect greater mindful qualities.
  ESRQ - 27 items, each scored 0-4, range 0-108, higher scores mean higher emotion regulation. Total scores used, no subscales. Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) has a range of scores from 12 to 48, each of the 12 items is rated on a 4-point Likert scale (from "Rarely/Not at all" to "Almost Always") with higher scores indicating greater mindfulness.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 9 | 10
units on a scale | -0.08 [-0.44 to 0.28] | 0.06 [-0.31 to 0.44]

10. Secondary Outcome: Physical Symptom Burden
Description: as for outcome 6
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver | Youth
Number analyzed (Participants) | 9 | 10
units on a scale | 7 [-19 to 33] | -3.5 [-16.4 to 9.4]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Caregiver | Youth
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT05241314/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT05241314/ICF_001.pdf